CLINICAL TRIAL: NCT03689751
Title: PIVOT: Patient Information Videos on Operations Trial. Patient Information Delivery for the Elective Preoperative Patient; A Single Blinded Randomised Controlled Trial
Brief Title: Patient Information Videos on Operations Trial
Acronym: PIVOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1210701
Record Dates: First submitted 2018-09-07; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Patient Education
Keywords: multimedia

STUDY DESIGN:
Intervention Model Description: Two RSAV were created explaining LSCS and TVT/TOT. Participants were block-randomised in groups of 10 to either control (no video) or intervention (video). Target recruitment was 60 patients per group; 30 patients per arm.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients were block randomised in groups of 10 participants to either control (no video) or intervention (video), using opaque envelopes. Both control and intervention arms received standard pre-operative face to face counseling and written information. Clinicians were blinded to allocation. A research nurse blinded to allocation performed data entry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LSCS Control Arm (No Intervention): Patients undergoing elective LSCS allocated to this arm underwent the normal preoperative educational pathway. This typically included face-to-face consultation and written information leaflets.
- LSCS Intervention ArmIntervention Arm (Experimental): Patients undergoing elective LSCS allocated to this arm underwent the normal preoperative educational pathway, but prior to the operation were shown the educational RSAV (LSCS Video) as an additional educational resource.
  Interventions: Other: LSCS Video
- TVT/TOT Control Arm (No Intervention): Patients undergoing elective TVT/TOT allocated to this arm underwent the normal preoperative educational pathway. This typically included face-to-face consultation and written information leaflets.
- TVT/TOT Interventional Arm (Experimental): Patients undergoing elective TVT/TOT allocated to this arm underwent the normal preoperative educational pathway, but prior to the operation were shown the educational RSAV (TVT/TOT Video) as an additional educational resource.
  Interventions: Other: TVT/TOT Video

INTERVENTIONS:
Other: LSCS Video — LSCS video created depicting the patient journey for elective LSCS patients.
  Arms: LSCS Intervention ArmIntervention Arm
Other: TVT/TOT Video — TVT/TOT video created depicting the patient journey for elective TVT/TOT patients.
  Arms: TVT/TOT Interventional Arm

SUMMARY:
This study evaluates whether rapid sequence animation videos (RSAV) are of use as an additional learning resource for the elective pre-operative patient. The investigators aimed to do this by comparing the change in knowledge and anxiety in two groups; Half of the patients were allocated to the normal patient pathway and the other half received the educational video as an additional preoperative learning resource.

DETAILED DESCRIPTION:
This single centre single-blinded randomised controlled study evaluates whether rapid sequence animation videos (RSAV) are of use as an additional learning resource for the elective pre-operative patient. The investigators aimed to do this by comparing the change in knowledge and anxiety from baseline to immediately preoperatively. Patients were block randomised to either the normal patient pathway or to receive the educational video as an additional preoperative learning resource.

Patients over 18 years of age electively listed for lower segment caesarean section (LSCS) and transobturator / transvaginal tape (TVT/TOT) were included.

Two RSAV were created explaining LSCS and TVT/TOT. Participants were block-randomised in groups of 10 to either control (no video) or intervention (video). Two questionnaires assessing anxiety were completed at baseline and immediately preoperatively using a Visual Analogue Scale (VAS) and a State- Trait Anxiety Inventory (STAI). Patient knowledge was assessed using a custom questionnaire. Primary outcome measures were the change in knowledge and anxiety scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients due to have one of the following operations: Elective Caesarean Section, Trans-Vaginal / Trans-Obturator Tape
* Patients must be consented for the operation before participating in stage 2 of the study.
* English speaking

Exclusion Criteria:

* Any conditions which may affect capacity: eg dementia, previous CVE or reduced cognitive ability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety from baseline to immediately preoperatively using a Visual Analogue Scale | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  Change in Anxiety from baseline to immediately preoperatively using a Visual Analogue Scale (VAS). This will be assessed using questionnaires, of which two will be completed: at baseline (stage 1) and immediately preoperatively (stage 2).
  VAS is a ten point linear scale where participants mark the corresponding value for their level of anxiety, where 0 is 'no anxiety' and 10 is 'extremely anxious'. Change will be recorded as points scored immediately preoperatively (stage 2) minus baseline score (stage 1), and referred to as an absolute number. An overall reduction in anxiety is therefore a negative integer, while an increase in anxiety is a positive integer.
Change in Knowledge from baseline to immediately preoperatively using a customised questionnaire where patients self-rated their knowledge related to the operation or condition. | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  Change in Knowledge from baseline to immediately preoperatively using a customised questionnaire where patients self-rated their knowledge related to the operation or condition. Each question has a ten-point scale, where the 0 points is 'not at all informed' and 10 points is 'extremely well informed'. Total scores are converted to a percentage (the higher percentage equating to being better informed) and change calculated as score at stage 2 minus score at stage 1. A negative percentage score for change in knowledge would therefore be interpreted as a reduction in knowledge, and a positive percentage score would be an increase in knowledge over the given time. The higher the change in percentage score, the bigger the change in knowledge noted by the participant.
Change in Anxiety from baseline to immediately preoperatively using the State-Trait Anxiety inventory (STAI) | From baseline at preoperative assessment to immediately preoperatively: 24 hours.
  Change in Anxiety from baseline to immediately preoperatively using the State-Trait Anxiety inventory (STAI).This will be assessed using questionnaires, of which two will be completed: at baseline (stage 1) and immediately preoperatively (stage 2). STAI is a validated anxiety score with a maximum score of 80 (extremely anxious) and minimum score of 20 (not at all anxious). These scores are converted to percentages, so 0% is not at all anxious, and 100% is extremely anxious.
  Change will be recorded as points scored immediately preoperatively (stage 2) minus baseline score (stage 1). Therefore a negative percentage score for change in anxiety measured by STAI equates to a reduction in anxiety, whilst a positive percentage change in anxiety measured by STAI equates to an increase in anxiety during the given time.

SECONDARY OUTCOMES:
Recruitment rate over the study period | Through study completion. This will assess enrolment rate. Number of participants approached and number of participants enrolled will be recorded throughout the study recruitment period of 18 months.
  Assess the recruitment rate for each group

CONTACTS AND LOCATIONS:
Overall Officials: Myles Taylor, BMBCh PhD, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient information data may be made available on individual request. Final study report and results summary will be freely available.

REFERENCES:
- See also: LSCS Project — https://youtu.be/E4qIAhFOcGk
- See also: PIVOT TVT/TOT — https://www.youtube.com/watch?v=sye-KPqcJhU

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03689751/Prot_SAP_ICF_000.pdf